CLINICAL TRIAL: NCT06155552
Title: Exploring Enrollment and Participation Patterns in Weight Loss Clinical Trials Patients: An Observational Clinical Trial Perspective
Brief Title: Evaluating the Occurrence of Participation Trends Among Weight Loss Clinical Trials Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 66708946
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Weight Loss
Keywords: weight loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical studies, with a distinct focus on weight loss, play a crucial role in evaluating the safety and effectiveness of novel treatments. These trials serve as instrumental means to determine whether new medications surpass conventional therapies, providing substantial evidence for their broader adoption.

The primary objective is to meticulously scrutinize trial completion rates and voluntary withdrawals within this specific patient group.

ELIGIBILITY:
Inclusion Criteria:

* Interested in losing weight and not enrolled in a formal weight loss program or taking medications or supplements that may cause weight change
* Participant must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study.
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed

Exclusion Criteria:

* Enrolled in another research study
* Inability to provide written informed consent
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Weight loss clinical trials patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a weight loss clinical study. | 3 months
Number of weight loss study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sarma S, Palcu P. Weight loss between glucagon-like peptide-1 receptor agonists and bariatric surgery in adults with obesity: A systematic review and meta-analysis. Obesity (Silver Spring). 2022 Nov;30(11):2111-2121. doi: 10.1002/oby.23563. PMID 36321278
- [Background] Palacios OM, Kramer M, Maki KC. Diet and prevention of type 2 diabetes mellitus: beyond weight loss and exercise. Expert Rev Endocrinol Metab. 2019 Jan;14(1):1-12. doi: 10.1080/17446651.2019.1554430. Epub 2018 Dec 6. PMID 30521416
- [Background] Jin S, Lu Q, Sun Y, Xiao S, Zheng B, Pang D, Yang P. Nutrition impact symptoms and weight loss in head and neck cancer during radiotherapy: a longitudinal study. BMJ Support Palliat Care. 2021 Mar;11(1):17-24. doi: 10.1136/bmjspcare-2019-002077. Epub 2020 Feb 4. PMID 32019753

DOCUMENTS (1):
  • Informed Consent Form (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT06155552/ICF_000.pdf